CLINICAL TRIAL: NCT02288897
Title: PV-10 Intralesional Injection vs Systemic Chemotherapy or Oncolytic Viral Therapy for Treatment of Locally Advanced Cutaneous Melanoma
Brief Title: PV-10 vs Chemotherapy or Oncolytic Viral Therapy for Treatment of Locally Advanced Cutaneous Melanoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inadequate rate of enrollment
Sponsor: Provectus Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Provectus Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PV-10-MM-31
Record Dates: First submitted 2014-11-04; First posted 2014-11-11 (Estimated); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Cutaneous Melanoma
Keywords: Stage III; Stage IIIB; Stage IIIC; Stage IV (M1a); Stage 3; Stage 4; IVM1a; IV(M1a); IV-M1a; in-transit; in transit; intransit; satellite; recurrent
MeSH Terms: conditions — Melanoma; Recurrence | interventions — Rose Bengal; Dacarbazine; Temozolomide; talimogene laherparepvec

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded review by independent review committee (IRC) for primary and key secondary endpoints.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PV-10 (Experimental): Subjects will receive intralesional PV-10 to all Study Lesions on study Day 1. PV-10 should be re-administered at 28-day intervals until complete response, disease progression or study termination occurs.
  Interventions: Drug: PV-10 (10% rose bengal disodium)
- Chemotherapy or Oncolytic Viral Therapy (Active Comparator): Subjects will receive (a) dacarbazine (intravenously at 850 m/m2) or temozolomide (orally at 200 mg/m2 daily for 5 consecutive days), administered at consecutive 28-day intervals, or (b) intralesional talimogene laherparepvec administered on an initial 21 interval followed by consecutive 14 day intervals, until complete response, disease progression or study termination occurs.
  Interventions: Drug: Dacarbazine, temozolomide or talimogene laherparepvec

INTERVENTIONS:
Drug: PV-10 (10% rose bengal disodium)
  Arms: PV-10
Drug: Dacarbazine, temozolomide or talimogene laherparepvec
  Arms: Chemotherapy or Oncolytic Viral Therapy

SUMMARY:
This is an international multicenter, open-label, randomized controlled trial (RCT) of single-agent intralesional PV-10 versus systemic chemotherapy or intralesional oncolytic viral therapy to assess treatment of locally advanced cutaneous melanoma in patients who (1) are not candidates for targeted therapy and (2) are not candidates for an immune checkpoint inhibitor. Subjects in the comparator arm will receive the Investigator's choice of dacarbazine (DTIC), temozolomide (TMZ) or intralesional talimogene laherparepvec as determined by Investigator preference and standard of care in the Investigator's country or region. Effectiveness will be assessed by comparison of progression-free survival (PFS) between all intent-to-treat (ITT) subjects in the two study treatment arms.

DETAILED DESCRIPTION:
Subjects will be randomized using a 2:1 treatment allocation (i.e. two-thirds of the subjects will receive PV-10).

Subjects in the comparator arm who have completed at least 1 cycle of study treatment and who meet the study protocol definition of disease progression but do not have evidence of visceral metastases will be eligible to enter the crossover portion of the study and receive PV-10. Subjects crossing over must meet all study inclusion and exclusion criteria for clinical laboratories, thyroid function, concurrent or intercurrent illness and pregnancy at the time of crossover.

Assessment of progression will be performed by an Independent Review Committee (IRC) based on Response Evaluation Criteria in Solid Tumors (RECIST) ver. 1.1 criteria. Events signaling progression include increase in size and/or number of lesions, distant or nodal disease progression, or death. All secondary endpoints involving disease response and progression will be based on the IRC determination.

An interim assessment of efficacy and safety will be performed by the IRC when 50% of the events required for the primary endpoint have occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, male or female
2. Histologically or cytologically confirmed melanoma
3. Recurrent, satellite or in-transit locally advanced cutaneous or subcutaneous melanoma metastases (i.e., American Joint Committee on Cancer (AJCC) Stage IIIB, IIIC or Stage IV M1a with no active nodal metastases)
4. At least 1 measurable Target Lesion that can be accurately measured by calipers or computed tomography (CT) consisting of:

   * at least one cutaneous lesion (each lesion ≥ 10 mm in longest diameter or up to 5 lesions having a sum of longest diameters ≥ 10 mm); and/or
   * at least one subcutaneous lesion (each lesion ≥ 10 mm in longest diameter by CT);
   * where Target Lesions should be at least 10 mm from any other lesion
5. No lesion > 50 mm in longest diameter; and no more than 50 lesions
6. Calculated required PV-10 dose ≤ 15 mL (based on total tumor burden)
7. Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-2
8. Not a candidate for treatment with an immune checkpoint inhibitor (e.g., failed or did not tolerate prior therapy, or due to co-morbidities, pre-existing autoimmune disease, drug unavailability or standard of care)
9. Not a candidate for targeted therapy with BRAF or combined BRAF/MEK inhibitors (e.g., failed or did not tolerate prior therapy, BRAF V600 wild-type or due to drug unavailability or standard of care)
10. Clinical Laboratories:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L and platelet count ≥100 x 10^9/L
    * Creatinine ≤ 3 times the upper limit of normal (ULN)
    * Estimated creatinine clearance (CrCl) or estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2
    * Total bilirubin ≤ 3 times the upper limit of normal (ULN)
    * Aspartate transaminase (AST), alanine transaminase (ALT) and alkaline phosphatase (ALP) ≤ 5 times the upper limit of normal (ULN)
    * Lactate dehydrogenase (LDH) ≤ 2 times the upper limit of normal (ULN).
11. Thyroid function abnormality ≤ Grade 2
12. Candidate for at least one comparator drug:

    * Subjects must be candidates for at least one of the designated comparator drugs

Exclusion Criteria:

1. Presence or history of visceral melanoma metastasis
2. Presence of active nodal metastases (e.g., radiologic or clinical evidence of current nodal disease)
3. Presence of more than 50 melanoma lesions
4. Radiation therapy to any Study Lesion within 6 weeks of initial study treatment.
5. Chemotherapy or other systemic cancer therapy within 4 weeks of initial study treatment (6 weeks for nitrosoureas or mitomycin), or regional chemotherapy (limb infusion or perfusion) within 12 weeks of initial study treatment
6. Immunotherapy for cancer within 4 weeks of initial study treatment
7. Local treatment (e.g., surgery, cryotherapy, laser ablation) to any Study Lesion within 4 weeks of initial study treatment
8. Anti-tumor vaccine therapy within 6 weeks of initial study treatment.
9. Investigational agents within 4 weeks of initial study treatment.
10. Concurrent or Intercurrent Illness:

    * Impaired wound healing or other extremity complications due to diabetes mellitus in subjects whose Study Lesions are located in an extremity
    * Severe peripheral vascular disease in subjects whose Study Lesions are located in an extremity
    * Significant concurrent or intercurrent illness, psychiatric disorders, or alcohol or chemical dependence that would, in the opinion of the Investigator, compromise the subject's safety or compliance or interfere with interpretation of study results.
    * Uncontrolled thyroid disease or cystic fibrosis
    * Clinically significant acute or unstable cardiovascular, cerebrovascular (stroke), renal, gastrointestinal, pulmonary, immunological, endocrine, or central nervous system disorders
11. Pregnancy:

    * Female subjects who are pregnant or lactating
    * Female subjects who have positive serum pregnancy test taken within 14 days of study treatment
    * Female subjects of child-bearing potential who are unwilling to use highly effective contraception (e.g., combined (estrogen and progestogen containing) or progestogen-only hormonal contraceptives, intrauterine devices, bilateral tubal ligation, vasectomized partner, sexual abstinence or equivalent measures) for the duration of study treatment
12. Contraindication for all comparators:

    * Subjects with contraindications to all of the designated comparator drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wachter, Ph.D., Study Director — Provectus Biopharmaceuticals, Inc.; Sanjiv Agarwala, M.D., Principal Investigator — St Luke's University Hospital and Health Network
Locations (23):
- United States (12):
  - Sharp Memorial Hospital - Clinical Oncology Research, San Diego, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Washington University School of Medicine - Dermatology, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Atlantic Health System, Morristown, New Jersey
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - St Luke's University Hospital and Health Network, Easton, Pennsylvania
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - M.D. Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- France (2):
  - Unité Cancéro-Dermatologie, Hôtel-Dieu CHU Nantes, Nantes
  - Institut Claudius Regaud, IUCT ONCOPOLE, Toulouse
- Germany (4):
  - Klinik für Dermatologie, Venerologie und Allergologie Charite Universitätsmedizin Berlin, Berlin
  - Klinik für Dermatologie Universitätsklinikum Essen Studienzentrum, Essen
  - Klinik für Dermatologie, Venerologie und Allergologie Universitätsklinikum Schleswig-Holstein Hautkrebszentrum, Kiel
  - Hautklinik Klinikum der Johannes Gutenberg Universität Hautkrebszentrum, Mainz
- Italy (3):
  - IRCCS Instituto Nazionale Tumori "Fondazione Giovanni Pascale", Napoli
  - Istituto Dermopatico dell'Immacolata (IDI IRCCS), Rome
  - Azienda Sanitaria Azienda Ospedaliera Universitaria Senese, Siena
- Mexico (2):
  - Centro de Estudios y Prevención del Cancer A.C., Juchitán de Zaragoza, Oaxaca
  - Neurociencias Estudios Clínicos S.C., Culiacán, Sinaloa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment open: Apr 2015; first patient treated: Nov 2015; last patient visit completed: Apr 2019
Groups:
- PV-10 (10% Rose Bengal Disodium): Subjects received intralesional PV-10 to all Study Lesions on study Day 1. PV-10 was re-administered at 28-day intervals until complete response, disease progression or study termination.
- Chemotherapy or Oncolytic Viral Therapy (Dacarbazine, Temozolomide or Talimogene Laherparepvec): Subjects received (a) dacarbazine (intravenously at 850 m/m2) or temozolomide (orally at 200 mg/m2 daily for 5 consecutive days), administered at consecutive 28-day intervals, or (b) intralesional talimogene laherparepvec administered on an initial 21 interval followed by consecutive 14 day intervals, until complete response, disease progression or study termination.
Period: Overall Study
Arm/Group | PV-10 (10% Rose Bengal Disodium) | Chemotherapy or Oncolytic Viral Therapy (Dacarbazine, Temozolomide or Talimogene Laherparepvec)
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PV-10: Subjects received intralesional PV-10 to all Study Lesions on study Day 1. PV-10 was re-administered at 28-day intervals until complete response, disease progression or study termination.
- Chemotherapy or Oncolytic Viral Therapy: Subjects received (a) dacarbazine (intravenously at 850 m/m2) or temozolomide (orally at 200 mg/m2 daily for 5 consecutive days), administered at consecutive 28-day intervals, or (b) intralesional talimogene laherparepvec administered on an initial 21 interval followed by consecutive 14 day intervals, until complete response, disease progression or study termination.
- Total: Total of all reporting groups
Arm/Group | PV-10 | Chemotherapy or Oncolytic Viral Therapy | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 9 | 3 | 12
Age, Continuous [Median (Full Range); unit: years] | 79.0 [47 to 90] | 66.8 [43 to 80] | 71.5 [43 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 7 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16
  Italy | 3 | 0 | 3
  France | 0 | 1 | 1
American Joint Committee on Cancer (AJCC) Stage at Baseline [Count of Participants; unit: Participants] — Disease burden was assessed at baseline to characterize melanoma disease stage according to the AJCC 2009 staging system, where stage (I-IV) is based on TNM classification: T refers to tumor size, N refers to lymph node involvement, and M represents metastasis (spread) to other parts of the body. The staging number represents a sum of the TNM classification: a lower stage (i.e., I or II) represents better the prognosis for the patient; the higher the stage (i.e., III or IV), the worse the prognosis.
  Participants were not stratified according to stage.
  Participants
    IIIB-IIID | 10 | 7 | 17
    IV-M1a | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was estimated via Kaplan-Meier analysis using Response Evaluation Criteria In Solid Tumors (RECIST v1.1) criteria. Subjects who did not have an event of progression or death were censored at their last assessment date.
  Assessment of progression was performed by the sponsor based on review of lesion measurement and clinical progression data reported by each investigator. Events signaling progression included increase in size and/or number of study lesions, onset of visceral metastatic disease, and death. For target lesions (assigned prior to randomization), complete response (CR) required disappearance of all target lesions; partial response (PR) required >= 30% decrease in sum of the longest diameter (SLD) of all target lesions; progressive disease (PD) required >=20% increase in SLD of target lesions. Non-target lesions were followed for CR, PD, or non-CR/non-PD status using equivalent thresholds. Progression occurred when PD was observed in either target or non-target lesion.
Time Frame: Assessed every 12 weeks until disease progression, withdrawal of consent, or study termination; progression detected between formal assessments was documented at the time of detection; median follow-up time for PFS was 26.6 weeks, maximum was 125.8 weeks.
Population: Subjects receiving PV-10 upon crossover from comparator are not included in the analysis population.
  Response data from one study center were censored due to resignation of the principal investigator.
  Because the study was terminated prior to achievement of pre-specified efficacy thresholds (i.e., out of a planned 225 subjects only 20 initiated study treatment), the small number of subjects enrolled precludes scientifically meaningful interpretation of PFS.
Measure: Median (Full Range); unit: Months
Groups:
- PV-10: Subjects received intralesional PV-10 to all Study Lesions on study Day 1. PV-10 should be re-administered at 28-day intervals until complete response, disease progression or study termination.
Arm/Group | PV-10 | Chemotherapy or Oncolytic Viral Therapy
Number analyzed (Participants) | 9 | 6
Months | 6.1 [1.5 to 28.9] | 8.6 [1.8 to 14.4]

2. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR was assessed using RECIST v1.1 criteria, and required disappearance of all target and non-target lesions.
Time Frame: Assessed every 12 weeks until disease progression, withdrawal of consent, or study termination; median follow-up time for CRR was 26.6 weeks, maximum was 125.8 weeks.
Population: Subjects receiving PV-10 upon crossover from comparator are not included in the analysis population.
  Response data from one study center were censored due to resignation of the principal investigator.
  Because the study was terminated prior to achievement of pre-specified efficacy thresholds (i.e., out of a planned 225 subjects only 20 initiated study treatment), the small number of subjects enrolled precludes scientifically meaningful interpretation of CRR.
Measure: Count of Participants; unit: Participants
Arm/Group | PV-10 | Chemotherapy or Oncolytic Viral Therapy
Number analyzed (Participants) | 9 | 6
Participants | 3 | 2

3. Secondary Outcome: Duration of Complete Response (DCR)
Description: DCR was estimated via Kaplan-Meier analysis for participants achieving a complete response, and was defined as the interval from first complete response to disease progression or death; responders who did not have an event of progression or death were censored at their last assessment date. Complete response was assessed using RECIST v1.1 criteria, and required disappearance of all target and non-target lesions.
Time Frame: Assessed every 12 weeks until disease progression, withdrawal of consent, or study termination; median follow-up time for DCR was 26.7 weeks, maximum was 77.7 weeks.
Population: Subjects receiving PV-10 upon crossover from comparator are not included in the analysis population.
  Response data from one study center were censored due to resignation of the principal investigator.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PV-10 | Chemotherapy or Oncolytic Viral Therapy
Number analyzed (Participants) | 3 | 2
Months | NA [NA to NA] — Could not be estimated due to the low number of events (fewer than 50% of complete responders in the study arm experienced progression prior to study termination). | NA [NA to NA] — Could not be estimated due to the low number of events (fewer than 50% of complete responders in the study arm experienced progression prior to study termination).

4. Secondary Outcome: Overall Survival (OS)
Description: OS was documented at 12 week intervals commencing on withdrawal from active study participation. Documentation was made by subject clinic visit or other personal contact, telephonic contact, review of medical records, or other unequivocal evidence of survival status. OS was estimated via Kaplan-Meier analysis, and was defined as the interval from randomization to death; subjects who did not have an event of death were censored at their last assessment date.
Time Frame: Assessed every 12 weeks upon withdrawal from active study participation until death, withdrawal of consent, or study termination; median follow-up time for survival was 82.4 weeks, maximum was 167.0 weeks.
Population: Subjects were analyzed according to treatment group assignment at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PV-10 | Chemotherapy or Oncolytic Viral Therapy
Number analyzed (Participants) | 12 | 8
Months | NA [NA to NA] — Could not be estimated due to the low number of events (fewer than 50% of subjects in the study arm died from any cause prior to study termination). | NA [NA to NA] — Could not be estimated due to the low number of events (fewer than 50% of subjects in the study arm died from any cause prior to study termination).

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Safety and tolerability were assessed by monitoring the frequency, duration, severity and attribution of adverse events and evaluating changes in laboratory values and vital signs.
Time Frame: Assessed every 4 weeks until 28 days after last treatment; median duration of treatment was 11.8 and 9.5 weeks in each treatment group, respectively.
Population: PV-10 safety population includes two subjects who received PV-10 upon crossover after progression on comparator.
Measure: Count of Participants; unit: Participants
Arm/Group | PV-10 | Chemotherapy or Oncolytic Viral Therapy
Number analyzed (Participants) | 14 | 8
Participants | 14 | 8

6. Other Pre Specified Outcome: Change in Domain Scores From Baseline Using the Patient Reported Skindex-16 Instrument
Description: In this exploratory endpoint, changes in Skindex-16 self-assessment scores were evaluated vs Day 1 baseline domain scores: symptom domain (items 1-4); emotional domain (items 5-11); and functioning domain (items 12-16). The Skindex-16 instrument solicits response to the extent of bother during the preceding week by 16 items (e.g., itching, hurting, worry, impact on daily activities), using a score from 0 (never bothered) to 6 (always bothered) for each item. Item scores are transformed to 0 to 100 scale, and domain scores are calculated as the average of the item scores comprising the domain. A lower domain score at baseline signifies lower impact of that domain; a decrease in domain score from baseline signifies improvement in that domain. Median baseline score and change from baseline over the study interval is presented for each domain.
Time Frame: Assessed at baseline (Day 1 at start of study treatment) and at the end of each treatment cycle (every 4 or 6 weeks) until disease progression, withdrawal of consent, or study termination; median follow-up time was 26.6 weeks, maximum was 125.8 weeks.
Population: Subjects receiving PV-10 upon crossover from comparator are included in the analysis population for PV-10 (after crossover).
  Response data from one study center were censored due to resignation of the principal investigator.
  Because the study was terminated prior to achievement of pre-specified efficacy thresholds (i.e., out of a planned 225 subjects only 20 initiated study treatment), the small number of subjects enrolled precludes scientifically meaningful interpretation of Skindex data.
Measure: Median (Standard Error); unit: Scores on a Scale (0-100)
Arm/Group | PV-10 | Chemotherapy or Oncolytic Viral Therapy
Number analyzed (Participants) | 10 | 6
Scores on a Scale (0-100)
  Baseline Symptom Domain Score | 2.1 (9.4) | 18.8 (11.2)
  Change in Symptom Domain Score from Baseline | -2.1 (6.0) | -6.3 (10.9)
  Baseline Emotional Domain Score | 20.2 (7.4) | 16.7 (15.5)
  Change in Emotional Domain Score from Baseline | -10.1 (6.3) | -4.8 (19.9)
  Baseline Functioning Domain Score | 1.7 (7.4) | 8.3 (8.9)
  Change in Functioning Domain Score from Baseline | -1.7 (6.1) | 6.7 (11.0)

ADVERSE EVENTS:
Time Frame: All adverse events occurring between signing the informed consent form and 28 days following final administration of study drug, or that occurred at any time that might be at least possibly related to study drug, were followed until: 1. the event resolved; 2. the subject was lost to follow-up; 3. the event was otherwise explained; or 4. no further improvement or worsening was expected. Median duration of treatment was 11.8 and 9.5 weeks in each treatment group, respectively.
Groups:
- PV-10: Subjects received intralesional PV-10 to all Study Lesions on study Day 1. PV-10 should be re-administered at 28-day intervals until complete response, disease progression or study termination.
  PV-10 (10% rose bengal disodium)
  PV-10 safety population includes two subjects who received PV-10 upon crossover after progression on comparator
- Chemotherapy or Oncolytic Viral Therapy: Subjects received (a) dacarbazine (intravenously at 850 m/m2) or temozolomide (orally at 200 mg/m2 daily for 5 consecutive days), administered at consecutive 28-day intervals, or (b) intralesional talimogene laherparepvec administered on an initial 21 interval followed by consecutive 14 day intervals, until complete response, disease progression or study termination.
  Dacarbazine, temozolomide or talimogene laherparepvec
Arm/Group | PV-10 | Chemotherapy or Oncolytic Viral Therapy
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/8
Other Adverse Events (participants affected / at risk) | 13/14 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PV-10 (N=14) | Chemotherapy or Oncolytic Viral Therapy (N=8)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) — A subject receiving oncolytic viral therapy experienced Grade 3 glomerulonephritis manifest as elevated creatinine commencing with the final dose of study drug and resolving to Grade 1 within 4 weeks; study treatment was discontinued permanently.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PV-10 (N=14) | Chemotherapy or Oncolytic Viral Therapy (N=8)
Injection site pain (General disorders) | 12 (12) | 1 (1)
Injection sit oedema (General disorders) | 7 (7) | 0 (0)
Injection site pruritus (General disorders) | 7 (7) | 0 (0)
Injection site discharge (General disorders) | 5 (5) | 1 (1)
Injection site erythema (General disorders) | 5 (5) | 0 (0)
Injection site discolouration (General disorders) | 4 (4) | 0 (0)
Injection site inflammation (General disorders) | 3 (3) | 0 (0)
Injection site ulcer (General disorders) | 3 (3) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)
Injection site infection (General disorders) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Lethargy (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 3 (3) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vision blurred (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Planned accrual was 225 subjects. However, due to slow accrual during a period of rapid change in global drug development for cutaneous melanoma, the study was terminated early after 20 subjects initiated study treatment. Because the study was terminated prior to achievement of pre-specified efficacy thresholds, the planned central independent review was not conducted and the small number of subjects precluded formal analysis and scientifically meaningful interpretation of efficacy parameters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT02288897/Prot_SAP_000.pdf